CLINICAL TRIAL: NCT01879514
Title: Study of Standardized Treatment of Integrative Medicine With the Severe IgA Nephropath
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Shanghai 6th People's Hospital (Other); RenJi Hospital (Other)
Responsible Party: Principal Investigator, yueyi deng, Director, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHDC12010114
Record Dates: First submitted 2013-03-25; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; Therapy of Chinese medicine
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Group (Experimental): Chinese Herb Prescription Granule, 6g, Bid, po. 48weeks plus prednisone, 0.5mg-1mg/kg·d, po. 48weeks
  Interventions: Drug: Chinese Herb Prescription Granule plus prednisone
- Placebo (Placebo Comparator): Placebo of Chinese Herb Prescription Granule, 6g, Bid, po. 48weeks plus prednisone, 0.5mg-1mg/kg•d, po. 48weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese Herb Prescription Granule plus prednisone — Chinese Herb Prescription Granule includes ZiBuGanShen Granule and BuShenTongLuo Granule
  Arms: Combination Group
Drug: Placebo — Placebo includes placebo of ZiBuGanShen Granule and placebo of BuShenTongLuo Granule
  Arms: Placebo

SUMMARY:
IgA nephropathy(IgAN) is the highest incidence of kidney pathology in the primary nephropathy. In terms of differences in prognosis, severe IgA nephropathy,one of the most main primary renal disease,could cause the uremia. It will be significant that early indicators of prognosis and early intervention can be normalized and the scientific criteria for judging the efficacy of great clinical can be established. The subject based on the past study,literature research and various treatment will take the method of multi-center, double-blind, randomized, control to investigate the standard treatment of severe IgA nephropathy. Otherwise the uniformity and objectivity of Traditional Chinese Medicine (TCM) will be improved by the standardization of TCM research based on the epidemiological investigation and statistical analysis. The subject will determine the efficacy of more sensitive biomarkers and establish more scientific criteria for judging the effect with the application of urine proteomics and metabolomics technologies in order to operate in the formation of the standardization program of the treatment of severe IgA nephropathy with the Integrative medicine of TCM.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed by renal biopsy and clinical examination as primary IgA nephropathy.
* Pathology:upon Lee's grade Ⅲ
* Age :18-60 years old.
* Gender and nationality are not limited
* Chronic Kidney Disease(CKD) Stage 3:（59 ml/min>GFR>30ml/min/1.73m2）
* 24-hour urine protein:≥1.0g.Informed consent

Exclusion Criteria:

* Patients within the past 3 months had received immunosuppressive agents or cytotoxic therapy is greater than 4 weeks
* Patients within the past 3 months who have received corticosteroids (prednisone or prednisolone) dose of more than 20mg / d up to 4 weeks
* Patients suffering from acute or rapidly progressive glomerulonephritis
* Patients continue with active hepatitis B and abnormal liver function tests transaminase
* Patients with a history of malignant tumor or malignancy, HIV infection, history of mental illness, acute central nervous system disorders, severe gastrointestinal disease, prohibiting the use of immunosuppressive agents
* Abnormal glucose metabolism, fasting blood glucose more than 6.2mmol/L
* Pregnancy or breast-feeding women
* Receiving other clinical trials
* Associated with other serious diseases and organ dysfunction
* Combined life-threatening complications such as severe infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | 12 months
  Evaluation of renal function indicators

SECONDARY OUTCOMES:
24 hours urine protein | 12 months
  Evaluate the therapeutic effect

CONTACTS AND LOCATIONS:
Overall Officials: YueYi Deng, PHD,MD, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Department of Nephrology,Longhua Hospital, Shanghai, China